CLINICAL TRIAL: NCT00442208
Title: An Open-Label, Randomized, Comparative 3-Way Cross-Over Study to Evaluate the Effect of Food on the 24-Hour Intragastric pH at Day 5 After Twice Daily Oral Administration of PN 200 (Omeprazole/Naproxen) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: POZEN (Industry)
Responsible Party: David Taylor, Pozen Inc.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PN200-105
Expanded Access: Available
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Healthy
Keywords: Healthy adults; Phase I
MeSH Terms: interventions — Isradipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: PN 200

SUMMARY:
Primary: To compare the pharmacodynamic efficacy of PN 200 in controlling intragastric pH (percent time pH> 4.0) following twice daily administration at different dosing times relative to food (30 or 60 minutes prior to food or taken togeterh with food) on Day 5.

DETAILED DESCRIPTION:
This study is designed to evaluate the effect of different dosing times of PN 200 relative to food on the intragastric pH profile of PN 200. PN 200 contains immediate release omeprazole, which may be subject to acid degradation in the stomach. Food is known to have a buffering effect on acid and therefore may result in less degradation of immediate release omeprazole. Alternatively, food may decrease the absorption of omeprazole in the duodenum. The relative magnitude of these effects is unknown. The data from this study will aid in choosing the optimal timing of PN dosing relative to food in future studies. The study is not blinded because the primary endpoint (intragastric pH) is a physiological variable not believed to be readily influenced by conscious or subconscious subject control.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-lactating, non-pregnant female subjects who are 18-55 years of age
2. Female subjects are eligible for participation in the study if they are of:

   * Non-childbearing potential (i.e., physiologically incapable of becoming pregnant); or,
   * Childbearing potential, have a negative pregnancy test (urine) at screening, and at least one of the following applies or is agreed to by the subject:

     * Female sterilization or sterilization of male partner; or,
     * Hormonal contraception by oral route, implant, injectable, vaginal ring; or,
     * Any intrauterine device (IUD) with published data showing that the lowest expected failure rate is less than 1% per year;
     * Double barrier method (2 physical barriers or 1 physical barrier plus spermicide); or
     * Any other method with published data showing that the lowest expected failure rate is less than 1% per year
3. Physical examination findings within normal limits for age
4. Able to understand and comply with study procedures required and able and willing to provide written informed consent prior to any study procedures being performed

Exclusion Criteria:

1. History of hypersensitivity, allergy or intolerance to omeprazole or other proton-pump inhibitors
2. History of hypersensitivity, allergy or intolerance to any NSAID (including aspirin) and/or a history of NSAID-induced symptoms of asthma, rhinitis, and/or nasal polyps
3. History of peptic ulcer disease or other acid related gastrointestinal symptoms
4. Participation in any study of an investigational treatment in the 4 weeks before screening or participation in another study at any time during the period of this study
5. Any significant medical illness that would contraindicate participation in the study
6. Gastrointestinal disorder or surgery leading to impaired drug absorption
7. Any significant mental illness, such as schizophrenia or bipolar disorder
8. Cardio- or cerebrovascular disease, based on history or risk factors, or clinically significant ECG in the investigator's opinion
9. Personal or family history of an inherited or acquired bleeding disorder
10. Positive test result for H pylori at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24
Dates: Start 2007-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
To compare the pharmacodynamic efficacy of PN 200 in controlling intragastric pH (percent time pH > 4.0)

SECONDARY OUTCOMES:
To evaluate the effect of different dosing times of PN 200 on the pharmacokinetic properties of omeprazole

CONTACTS AND LOCATIONS:
Overall Officials: David Taylor, Study Director — POZEN
Locations (1):
- Pozen Inc., Chapel Hill, North Carolina, United States